CLINICAL TRIAL: NCT02461355
Title: Enhancing Aphasia Therapy With Anodal Transcranial Direct Current Stimulation in Chronic Stroke Patients
Brief Title: Transcranial Direct Current Stimulation for Post-Stroke Aphasia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Columbia University (Other)
Collaborators: Pitkin Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAO1700
Record Dates: First submitted 2015-04-08; First posted 2015-06-03 (Estimated); Results first posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anodal tDCS (Experimental): Anodal tDCS over the left posterior language areas during aphasia therapy for 8 one-hour sessions
  Interventions: Behavioral: Aphasia therapy; Device: Anodal tDCS
- Sham tDCS (Sham Comparator): Sham tDCS over the left posterior language areas during aphasia therapy for 8 one-hour sessions
  Interventions: Behavioral: Aphasia therapy; Device: Sham tDCS

INTERVENTIONS:
Behavioral: Aphasia therapy — Aphasia therapy using a computerized scripting program
Device: Anodal tDCS — Anodal transcranial direct current stimulation using the Chattanooga Ionto device
  Arms: Anodal tDCS
Device: Sham tDCS — Sham transcranial direct current stimulation using the Chattanooga Ionto device
  Arms: Sham tDCS

SUMMARY:
This is a randomized, crossover design trial that will compare how anodal transcranial direct current stimulation (tDCS) versus sham tDCS administered during multiple sessions of scripting therapy affects the acquisition and retention of trained scripts.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 21 years
2. Ischemic left hemispheric stroke verified by imaging (CT or MRI) greater than 6 months ago
3. Residual non-fluent or anomic aphasia, with Western Aphasia Battery-Revised Aphasia Quotient score <60
4. Fluent English speaker prior to stroke
5. Right-handed prior to stroke
6. Ability to give informed consent and understand the tasks involved.

Exclusion Criteria:

1. History of recurrent stroke, either ischemic or hemorrhagic, in the left middle cerebral artery territory
2. Imaging unavailable
3. Large middle cerebral artery infarct involving entire inferior division (temporo-parietal) territory
4. History of dementia prior to the stroke
5. History of seizure, prior electroconvulsive therapy, deep brain stimulators, or brain surgery
6. Social and/or personal circumstances that interfere with ability to return for therapy and assessment sessions.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomoko Kitago, MD, Principal Investigator — Columbia University
Locations (1):
- Adler Aphasia Center, Maywood, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Includes participants who received anodal transcranial direct current stimulation (tDCS) or sham tDCS over the left posterior language areas during aphasia therapy for 8 one-hour sessions.Since the PI left the institution and data on the cross-over assignment is not available for the 2 participants, data was reported on the collective whole and not on the treatment assignment per individual.
Period: Overall Study
Arm/Group | All Participants
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Includes participants who received anodal transcranial direct current stimulation (tDCS) or sham tDCS over the left posterior language areas during aphasia therapy for 8 one-hour sessions.
Arm/Group | All Participants
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Correct of Trained Scripts
Time Frame: From Baseline to up to 2 days post-training
Population: Due to poor enrollment, data collection was not complete and therefore data was not analyzed. PI is now no longer at the institution.
Groups:
- All Participants: Includes participants who received anodal tDCS or sham tDCS over the left posterior language areas during aphasia therapy for 8 one-hour sessions.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Words Per Minute of Trained Scripts
Time Frame: From Baseline to up to 2 days post-training
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Percent Correct of Trained Scripts
Time Frame: Baseline to 2 weeks and 4 weeks post-training
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Words Per Minute of Trained Scripts
Time Frame: Baseline to 2 weeks and 4 weeks post-training
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Change in Percent Script Words Omitted
Time Frame: Baseline to immediate, 2 weeks, and 4 weeks post-training
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes